CLINICAL TRIAL: NCT06526247
Title: Evaluating Interventions for Intimate Partner Violence Use in Washington State
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Office of Crime Victims Advocacy - Washington State Department of Commerce (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-44938
Record Dates: First submitted 2024-07-25; First posted 2024-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Intimate Partner Violence
Keywords: Strength at Home (SAH); Trauma-informed; Treatment as Usual (TAU); Posttraumatic stress disorder (PTSD); Alcohol use; Washington state
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcohol Drinking | interventions — Therapeutics; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Intervention Model Description: Single site, controlled trial. All participants will be randomized at the individual level to SAH or TAU, with a 1:1 allocation ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength at Home (SAH) (Experimental): Participants randomized into this arm with receive a trauma-informed intimate partner violence (IPV) intervention program.
  Interventions: Behavioral: Strength at Home (SAH)
- Treatment as Usual (TAU) (Active Comparator): Participants randomized into this arm with receive a standard IPV intervention program in the state of Washington.
  Interventions: Behavioral: Treatment as usual for IPV

INTERVENTIONS:
Behavioral: Strength at Home (SAH) — SAH is a group intervention that incorporates elements from interventions for violence and trauma. It is administered during 12 two-hour weekly sessions. The program uses a social information processing model based on the premise that trauma negatively impacts one's ability to interpret and respond to social situations effectively. It underscores the importance of cognitive behavioral strategies to monitor one's thoughts and responses to interpersonal situations.
  Arms: Strength at Home (SAH)
Behavioral: Treatment as usual for IPV — Treatment as usual for IPV includes court-mandated interventions delivered over the 26 two-hour weekly sessions in Washington state.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Intimate partner violence (IPV), specifically physical and psychological aggression toward an intimate partner, represents a public health crisis that affects millions of Americans each year. There currently exists very little evidence from randomized controlled trials for the effectiveness of abuser intervention programs designed to prevent and end perpetration of IPV in the general population. This is troubling considering that approximately half a million men and women are court-mandated to these programs each year.

The investigators will conduct a randomized control trial (RCT) investigating the efficacy of the Strength at Home (SAH) intervention in reducing intimate partner violence (IPV). The overarching aim of this study is to test the efficacy of SAH with court-involved-partner-violent men through an RCT comparing those who receive SAH with those who receive other standard IPV interventions offered in the state of Washington (treatment as usual- TAU).

The specific aims are:

1.1: Compare the frequency of physical and psychological IPV, the primary outcomes of interest, across conditions as reported by the male participants and their intimate partners across Time 1 (baseline) and four 3-month follow ups (Times 2-5). It is expected that greater reductions in IPV frequencies will be evidenced in SAH than TAU over the course of the year.

1.2: Compare symptoms of PTSD, alexithymia, and alcohol use problems across conditions and assessment time points as reported by the male participants. It is expected that greater reductions in these symptoms will be evidenced in SAH than TAU over the course of the year.

1.3: Compare treatment satisfaction across conditions as reported by the male participants across the four 3-month follow ups (Times 2-5). It is expected that treatment satisfaction will be higher in SAH than TAU.

ELIGIBILITY:
Inclusion Criteria:

Men:

1. Identify as a man
2. Provide consent for the research team to contact his intimate partner(s) for data collection purposes;
3. Court-referred for IPV intervention in Washington state

Women:

1. Identify as a woman
2. Were or currently are an intimate partner involved in an incident of IPV with a court-referred participant

Exclusion Criteria:

1. demonstrates active psychosis that may interfere with their ability to participate in group
2. expresses prominent suicidal or homicidal ideation that requires hospitalization
3. does not possess proficiency in spoken English
4. periods of incarceration after study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
IPV assessment | Baseline, 3 months, 6 months. 9 months, 12 months
  The revised Conflict Tactics Scales (CTS2), a 20-item instrument, will be used to assess IPV. The Physical Assault (12 items) and Psychological Aggression (8 items) subscales will be administered. Each of the 20 items is scored by the frequency of occurrence of the item with 8 choices 1-7 and 0.
Psychological IPV assessment | Baseline, 3 months, 6 months. 9 months, 12 months
  The 7-item Restrictive Engulfment subscale of the Multidimensional Measure of Emotional Abuse (MMEA) will be used as an additional measure of psychological IPV. Each item has 7 potential responses from 0=never to 6= more than 20 times. Scores can range from 0 to 42, with higher scores being associated with more psychological IPV.
Post Traumatic Stress Disorder (PTSD) symptoms | Baseline, 3 months, 6 months. 9 months, 12 months
  The 20-item PTSD Checklist for DSM 5 (PCL-5) will be used to assess PTSD symptoms. It is a self-report measure. Items are rated on a 5-point Likert scale [0 to 4] and summed. Scores range from 0 to 80 with higher scores associated with more PTSD symptoms. A total score of 33 or higher may indicate severe PTSD.
Alcohol use | Baseline, 3 months, 6 months. 9 months, 12 months
  The 10-item Alcohol Use Disorders Identification Test (AUDIT) will be used to assess problem drinking behavior over the past six months, with higher scores reflecting greater alcohol misuse.
Alexithymia assessment | Baseline, 3 months, 6 months. 9 months, 12 months
  The 20-itemToronto Alexithymia Scale (TAS-20) will be used to assess alexithymia. The TAS-20 uses cutoff scoring, with scores of 52-60 indicating possible alexithymia, and scores above 60 indicating alexithymia.

SECONDARY OUTCOMES:
Treatment Satisfaction | 3 months, 6 months. 9 months, 12 months
  Participants' satisfaction will be assessed with a 4-item measure used in a study conducted by the Treatment of Depression Collaborative Research Program.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Taft, PhD, Principal Investigator — BU School of Medicine and National Center for PTSD
Locations (1):
- BU Chobanian & Avedisian School of Medicine, Psychiatry, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No